CLINICAL TRIAL: NCT07046624
Title: Development of an Infusion Monitoring System to Prevent Phlebitis, Infiltration and Extravasation and Its Application in the Intensive Care Unit
Brief Title: Prevention of Phlebitis, Infiltration and Extravasation With Infusion Monitoring System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Fatma Aksoy, Principal Investigator, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025/34
Record Dates: First submitted 2025-06-10; First posted 2025-07-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Extravasation; Intensive Care Units (ICUs); Phlebitis; Infiltration
MeSH Terms: conditions — Phlebitis | interventions — Patient Care

STUDY DESIGN:
Intervention Model Description: The clinics included in the study will be divided into two groups: experimental and control.
Who Masked: Outcomes Assessor
Masking Description: In blinding the results, only the person performing the analysis will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Group where no intervention will be applied
  Interventions: Behavioral: Infusion monitoring system developed for use by nurses in patient care
- Experimental group (Experimental): The group to which the intervention will be applied
  Interventions: Behavioral: Infusion monitoring system developed for use by nurses in patient care

INTERVENTIONS:
Behavioral: Infusion monitoring system developed for use by nurses in patient care — In the experimental group, the frequency of complications will first be determined and an infusion monitoring system will be developed and used by nurses in patient care.

SUMMARY:
Peripheral venous catheter complications are conditions that are frequently seen in intensive care clinics and require nursing care. The most common complications are phlebitis, infiltration and extravasation. Nurses should take the necessary precautions to prevent these complications from developing.. Therefore, this planned thesis study aims to establish an infusion monitoring system and evaluate its effectiveness in early detection of complications related to peripheral intravenous catheters. The research is planned as a randomized controlled experimental study. The study will be conducted in Ordu State Hospital General Intensive Care Unit 1 and General Intensive Care Unit 3 clinics. The universe of the study will consist of patients receiving inpatient treatment in General Intensive Care Unit 1 and General Intensive Care Unit 3 clinics. The sample size will be determined by g-power analysis after a two-month preliminary follow-up. Data will be collected with the "Clinical Follow-up Form", "Patient Information Form", and "Complication Follow-up Form". The clinics included in the study will be divided into two groups as experimental and control groups. First, the frequency of complications will be determined in the experimental and control groups. Then, while the control group continues its routine protocol and applications, an infusion follow-up system will be developed in the experimental group and will be used by nurses in patient care. In the final stage, the frequency of peripheral venous catheter complications will be determined again. Data will be evaluated using the SPSS 22.0 package program at a significance level of p<0.05 and a confidence interval of 95%.

DETAILED DESCRIPTION:
Electronic monitoring systems can increase the quality of care and patient safety by enabling nurses to gain effective care and application techniques and preventing complications that may develop in patients. In addition, the integration of such technologies into clinical practices can enable nurses to act more consciously. This study can lead to the wider application of technology-based solutions in healthcare services by showing the effects of electronic monitoring systems in patient care and complication management in the scientific literature. Reductions in phlebitis, infiltration and extravasation rates improve clinical outcomes by increasing patient safety and increase the quality of life of patients. It is expected that costs will decrease with the increase in the quality of healthcare services and it is aimed to reduce the workload of nurses. Reductions in complication rates can increase the welfare of individuals by allowing patients to recover faster and shorten the duration of hospital stay. In addition, reductions in health-related complications can help reduce healthcare expenses and ease the financial burden of the state and individuals.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Receiving medication via peripheral intravenous catheter,
* Monitored daily for signs of phlebitis, infiltration and extravasation,
* Patients who can speak

Exclusion Criteria:

* Unconscious patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-11-08 (Estimated); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-07-08 (Estimated)

PRIMARY OUTCOMES:
Complication Follow-up Form | From enrollment to the end of treatment at 10 monts
  This form was developed by the investigators to enable the identification and evaluation of phlebitis, infiltration and extravasation complications. This form has no minimum and maximum score.

SECONDARY OUTCOMES:
Peripheral Edema Scale | From enrollment to the end of treatment at 10 monts
  It helps to diagnose the oedema developing in the patient. A minimum score of 1 and a maximum score of 4 is obtained from the oedema scale. The increase in the score indicates an increase in the degree of oedema and more unfavourable results.
Glasgow Coma Scale | From enrollment to the end of treatment at 10 monts
  This scale allows the patients' level of consciousness to be assessed. Minimum 3 points and maximum 15 points can be obtained from this scale. An increase in the score indicates that the level of consciousness is better, while a decrease in the score indicates that the level of consciousness has worsened.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Aksoy, MscN, Principal Investigator — Ordu University; Şule Bıyık Bayram, PhD, Study Director — Karadeniz Technical University

IPD SHARING:
Plan to Share IPD: Yes
I just want to share the title of the study. I want the method of the study to remain secret for now since the study is not completed.
Supporting Information: Study Protocol
Time Frame: It can start and be published 3 months after the results are published.
Access Criteria: The data obtained from the research can be accessed after being analyzed with a suitable statistical program and the results shared.

REFERENCES:
- See also: Remote patient monitoring: a comprehensive study — https://link.springer.com/article/10.1007/s12652-017-0598-x
- See also: Design and Development of Patient Monitoring System — https://iopscience.iop.org/article/10.1088/1757-899X/226/1/012094/meta

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT07046624/Prot_SAP_002.pdf
  • Informed Consent Form (2025-07-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT07046624/ICF_003.pdf